CLINICAL TRIAL: NCT03008226
Title: Post Market Evaluation of the 9mm Spiration Valve System in Patients With Severe Heterogeneous Emphysema
Brief Title: Spiration Valve System 9 mm European Post Market Evaluation Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Collaborators: Lung Clinic Hemer (Other); Asklepios Kliniken Hamburg GmbH (Other); Otto Wagner Hospital (Other)
Responsible Party: Principal Investigator, Felix JF Herth, Prof. Dr. med., Heidelberg University
Other Study IDs: TKSPI 001/2014
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Implementation of 9 mm intrabronchial valves

SUMMARY:
The purpose of this observational study is to investigate the efficacy of 9 mm intrabronchial valve treatment in patients with heterogeneous emphysema and to gain further insights and experience on the treatment with this valve size.

DETAILED DESCRIPTION:
This study is designed to evaluate performance of the 9 mm valve system in patients with at least one airway to be treated . Patients with severe airflow obstruction, severe emphysema, significant hyperinflation, and moderate to severe dyspnea are eligible to be evaluated for enrollment in this study. In this study, eligible patients will have severe emphysema in a target lobe with an intact fissure. Patients must be able to tolerate a flexible bronchoscopy procedure. After evaluation of all inclusion and exclusion criteria, with review of the CT data by the core laboratories, patients will be enrolled in the study. The indications for endoscopic reduction of pulmonary volume with intrabronchial valves are presented in various preliminary examinations. The duration of the study is about 7 months for each patient. It involves an examination before the valves are inserted, the valves are inserted within the scope of a bronchoscopy, followed by a follow-up examination directly after the valves are inserted, a follow-up period of at least 3 nights in the appropriate clinic and follow-up visits 14, 30 each , 90 and 180 days after the valves are inserted.

The study is expected to enroll up to 30 patients who complete the 6 month follow-up visit at up to 4 sites with up to 15 patients per site.

ELIGIBILITY:
Inclusion Criteria:

* Patient is older than 40 years in age
* Patient has severe heterogeneous emphysema with moderate to severe dyspnea as defined as an mMRC of 2 or greater.
* The target lobe and ipsilateral lobe will be separated with an intact fissure, as determined by HRCT (> 90% integrity).
* Patient has received standard-of-care medical management and it has been stable for 6 weeks.
* Patient can walk a minimum of 140 meters in the six minute walk test.
* Patient's obstructive disease is severe as defined by: FEV1 ≤45% of predicted
* Patient's hyperinflation is defined by: RV ≥ 150% of predicted
* Patient is willing to participate in a study, complete the required follow-up visits, and maintain consistent nutrition and exercise habits during the study period

Exclusion Criteria:

* Patient does not have at least one airway with the intention to be treated with a 9 mm Spiration Valve based on a calibrated balloon sizing of the airway.
* Patient has co-existing major medical disease that will limit evaluation, participation, or follow-up in the study
* Patient is unable to provide informed consent
* Patient is not an appropriate candidate for or is unable to tolerate, flexible bronchoscopy procedures
* Patient has history of 4 or more hospitalizations for COPD exacerbation or respiratory infections in the past year and none have occurred in the 3 months prior to baseline testing.
* Patient has giant bulla (> 1/3 volume of lung)
* Patient has severe pulmonary hypertension.
* Patient has bronchiectasis
* Patient has evidence of systemic disease or neoplasia expected to compromise survival during the 6-month study period
* Patient has had prior lung volume reduction surgery, intra-bronchial valve therapy for emphysema, or major lung procedures (lobectomy or greater).
* Patient has demonstrated unwillingness or inability to complete screening or baseline data collection procedures.
* Patient participated in a study of an investigational drug or device within the past 30 days prior to participation in this study, or is currently participating in another clinical study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with severe airflow obstruction, severe emphysema, significant hyperinflation, and moderate to severe dyspnea . Eligible patients will have severe emphysema in a target lobe with an intact fissure
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-01 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Mean changes in target lobe volume | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Felix Herth, Prof.Dr.med., Principal Investigator — University Heidelberg
Locations (1):
- Thoraxklinik, University of Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No